CLINICAL TRIAL: NCT00056862
Title: Low Dose Peginterferon and Ribavirin Therapy for Patients With Chronic Hepatitis C Infected With Genotype 2 or 3
Brief Title: Low-Dose Peginterferon and Ribavirin to Treat Chronic Hepatitis C in Patients Infected With HCV Genotype 2 or 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030136; 03-DK-0136 (Other: NIH Clinical Center)
Record Dates: First submitted 2003-03-25; First posted 2003-03-25 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus; Antiviral Agents; Hemolysis; Neutropenia; Cirrhosis; Hemolytic Anemia; Viral Hepatitis; Ribavirin; Alfa Interferon; Pegylated Interferon; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C; Hemolysis; Neutropenia; Fibrosis; Anemia, Hemolytic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-dose pegIFN/standard-dose RBV (Experimental): Patients receive a lower dose of peginterferon alfa-2a (90 mcg per week) and standard dose of ribavirin (800 mg/d) for chronic hepatitis C, genotype 2/3, for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Standard-dose PegIFN/RBV (Active Comparator): Patients receive the standard, recommended doses of peginterferon alfa-2a (180 mcg per week) and ribavirin (800 mg/d) for chronic hepatitis c, genotype 2/3, for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 90 mcg/week
  Other Names: Pegasys
  Arms: Low-dose pegIFN/standard-dose RBV
Drug: Peginterferon alfa-2a — 180 mcg/week
  Other Names: Pegasys
  Arms: Standard-dose PegIFN/RBV
Drug: Ribavirin — 800 mg/day
  Other Names: Copegus

SUMMARY:
This study will examine the effectiveness of low-dose peginterferon and ribavirin therapy for certain patients with chronic hepatitis C-a liver disease that, in some patients, can progress to cirrhosis of the liver, liver cancer, and liver failure.

DETAILED DESCRIPTION:
Sixty patients with chronic hepatitis C infected with HCV genotype 2 or 3 will be treated using the combination of either low- or standard dose peginterferon and ribavirin for 24 weeks, with re-treatment using the standard doses and a longer duration (48 weeks) for those who do not respond to or relapse after initial low dose therapy.

Adult patients with chronic hepatitis C who have HCV genotype 2 or 3 and previously have not received anti-viral treatment will be given peginterferon alfa-2a (90 or 180 micrograms weekly by injection) and ribavirin (800 mg daily by mouth). Patients will be monitored at 2- to 4-week intervals for side effects, compliance, complete blood counts, liver biochemical tests and HCV RNA. Patients becoming HCV RNA negative by week 12 will be considered on-treatment responders, continue therapy to week 24, and be monitored thereafter for another 24 weeks. Patients who do not become HCV RNA negative by week 12 as well as patients who relapse after therapy will be retreated with 180 micrograms of peginterferon weekly and 800 mg of ribavirin for another 48 weeks.

The primary outcome will be sustained loss of HCV RNA at 24 weeks after low- or standard-dose combination therapy. Secondary outcomes include viral kinetics and side effects. Because of preliminary results in the initial 31 patients enrolled in this study, the dose of peginterferon was changed from 90 to 180 micrograms weekly for the remaining 29 patients to be enrolled, allowing for a direct comparison of efficacy, viral kinetics and side effects of standard- vs low-dose peginterferon therapy.

This study will evaluate the relative efficacy and safety of the standard versus lower doses of peginterferon with ribavirin in patients with chronic hepatitis C and HCV genotype 2 or 3.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age above 18 years, male or female.

Presence of anti-HCV in serum.

Positive HCV RNA determination in serum.

HCV genotype 2 or 3 as determined by Inno LiPa assay or by direct sequencing. Patients with mixed genotypes will not be eligible if they have genotypes other than 2 or 3.

Written informed consent.

EXCLUSION CRITERIA:

Previous treatment with interferon alpha or peginterferon.

Decompensated liver disease, as marked by bilirubin greater than 4 mg/dL, albumin less than 3.0 g/dL, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy.

Patients with ALT levels greater than 1000 U/L (greater than 25 times ULN) will not be enrolled but may be followed until three determinations are below this level.

Pregnancy or, in women of child-bearing potential or in spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicidal, or birth control pills, or an intrauterine device.

Significant systemic or major illnesses other than liver disease, including congestive heart failure, renal failure (creatinine clearance less than 50 ml/min), organ transplantation, serious psychiatric disease not controlled by psychotropic agents, and angina pectoris.

Evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.

Pre-existing, severe bone marrow compromise; anemia (hematocrit less than 30%), neutropenia (less than 1000 neutrophils/microliter) or thrombocytopenia (less than 70,000 cells/microliter).

History of hemolytic anemia.

Evidence of another form of liver disease in addition to hepatitis C (for example hepatitis B, autoimmune liver disease, Wilson's disease, alcoholic liver disease).

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous six months.

Evidence of hepatocellular carcinoma: either alfa-fetoprotein (AFP) levels greater than 50 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Clinical gout.

HIV infection.

Quiescent or active, serious autoimmune disease such as lupus erythematosus, ulcerative colitis, Crohn's disease or rheumatoid arthritis that in the opinion of the investigators might be exacerbated by therapy with alfa interferon.

The use of immunosuppressive medications, including corticosteroids in doses of 10 mg of prednisone or its equivalent and higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-03; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rotman Yaron, MD, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liang TJ, Rehermann B, Seeff LB, Hoofnagle JH. Pathogenesis, natural history, treatment, and prevention of hepatitis C. Ann Intern Med. 2000 Feb 15;132(4):296-305. doi: 10.7326/0003-4819-132-4-200002150-00008. PMID 10681285
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Neumann AU, Lam NP, Dahari H, Gretch DR, Wiley TE, Layden TJ, Perelson AS. Hepatitis C viral dynamics in vivo and the antiviral efficacy of interferon-alpha therapy. Science. 1998 Oct 2;282(5386):103-7. doi: 10.1126/science.282.5386.103. PMID 9756471
- [Result] Rotman Y, Borg BB, Soza A, Feld JJ, Modi AA, Loomba R, Lutchman G, Rivera E, Doo E, Ghany MG, Heller T, Neumann AU, Liang TJ, Hoofnagle JH. Low- and standard-dose peginterferon alfa-2a for chronic hepatitis C, genotype 2 or 3: efficacy, tolerability, viral kinetics and cytokine response. Aliment Pharmacol Ther. 2010 May;31(9):1018-27. doi: 10.1111/j.1365-2036.2010.04263.x. Epub 2010 Jan 16. PMID 20163377
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-DK-0136.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Dec 2003 and Dec 2004, 31 patients were enrolled into the low-dose group and were treated with peginterferon alfa-2a 90ug/week and ribavirin 400 mg/twice daily for 24 week. From Feb 2005, all subsequent patients were enrolled into a standard-dose group and treated for 24 weeks with the doses of the approved regimen.
Groups:
- Low Dose Group: All patients receive peginterferon alfa-2a and ribavirin for 24 weeks with measurements of HCV RNA, routine liver tests, complete blood counts and side effects at regular intervals during therapy. Arm A receives a lower dose of peginterferon (90 mcg per week) but standard, recommended dose of ribavirin for chronic hepatitis C, genotype 2 and 3.
- Standard Dose Group: All patients receive peginterferon alfa-2a and ribavirin for 24 weeks with measurements of HCV RNA, routine liver tests, complete blood counts and side effects at regular intervals during therapy. Arm B receives the standard, recommended dose of peginterferon (180 mcg per week) and standard, recommended dose of ribavirin for chronic hepatitis c, genotype 2 and 3.
Period: Overall Study
Arm/Group | Low Dose Group | Standard Dose Group
Started | 31 | 27
Completed | 30 | 27
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Group | Standard Dose Group | Total
Number analyzed (Participants) | 30 | 27 | 57
Age Continuous [Mean (Full Range); unit: years] | 48 [29 to 62] | 47 [26 to 69] | 48 [26 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 26 | 20 | 46
  Asian | 2 | 5 | 7
  Hispanic | 1 | 0 | 1
  African-American | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
ALT [Mean (Standard Deviation); unit: U/L] | 91 (69) | 97 (85) | 94 (77)
HCV RNA [Mean (Standard Deviation); unit: log IU/mL] | 6.3 (0.82) | 5.9 (1.02) | 6.1 (0.92)
Genotype [Number; unit: participants]
  HCV Genotype 2 | 21 | 13 | 34
  HCV Genotype 3 | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Virological Response (Intention to Treat)
Description: Virological response category. Sustained virological response (SVR) is defined as negative serum HCV RNA at least 6 months after the end of treatment. Non-response is defined as serum HCV RNA positivity on week 12 of treatment. Breakthrough/relapse is defined as HCV RNA becoming negative and subsequently positive on treatment or after treatment is stopped.
Time Frame: 6 months after stopping therapy
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Low Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 27
participants
  Sustained Virological Response (SVR) | 19 | 21
  Relapse/breakthrough | 7 | 2
  Nonresponse | 3 | 1
  Treatment stopped for adverse event | 0 | 3
  Lost to follow-up | 1 | 0

2. Secondary Outcome: First Phase Decline in Logarithm of HCV RNA Level
Description: The 1st phase decline is defined as the log difference between baseline HCV RNA level and the level on day 2 of treatment (see Neumann et al, Science, 1998).
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: logIU/mL
Arm/Group | Low Dose Group | Standard Dose Group
Number analyzed (Participants) | 28 | 23
logIU/mL | 1.15 (0.88) | 2.20 (1.14)
Statistical Analysis 1: Comparison: Low Dose Group vs Standard Dose Group; Null hypothesis: first phase decline in HCV RNA are the same for the two groups; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

3. Primary Outcome: Virological Response Category (Per Protocol)
Description: as for outcome 1
Time Frame: 6 months after therapy
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Low Dose Group | Standard Dose Group
Number analyzed (Participants) | 28 | 23
participants
  SVR | 19 | 20
  Relapse/breakthrough | 7 | 2
  Nonresponse | 2 | 1

4. Secondary Outcome: Slope of Second Phase Decline in HCV Levels
Description: The 2nd phase slope is defined as the slope of the logarithmic viral levels from week 1 to week 4 of treatment (see Neumann et al, Science, 1998).
Time Frame: day 7 to day 28
Measure: Mean (Standard Deviation); unit: logIU/mL
Arm/Group | Low Dose Group | Standard Dose Group
Number analyzed (Participants) | 28 | 23
logIU/mL | 1.14 (0.69) | 1.39 (0.64)
Statistical Analysis 1: Comparison: Low Dose Group vs Standard Dose Group; Null hypothesis: the second phase slopes of HCV RNA are the same for the two groups; Test type: Superiority or Other; p = 0.2, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Time to Negativity
Description: Time from treatment initiation to the first negative HCV RNA test during treatment
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 27
days | 42 [32 to 51] | 28 [19 to 37]
Statistical Analysis 1: Comparison: Low Dose Group vs Standard Dose Group; Null hypothesis: the time to negativity for the two groups are same; Test type: Superiority or Other; p = 0.047, Log Rank

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Low Dose Group | Standard Dose Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 3/27
Other Adverse Events (participants affected / at risk) | 2/30 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Group (N=30) | Standard Dose Group (N=27)
Melanoma and death (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mastoiditis complicated by myocardial infarction, heart failure, coronary bypass surgery and death (Cardiac disorders) | 0 (0) | 1 (1)
Heroin overdose leading to death (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Group (N=30) | Standard Dose Group (N=27)
Sarcoidosis development (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (off treatment), (Cardiac disorders) | 1 (1) | 0 (0)
Severe hemolysis requiring transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes